CLINICAL TRIAL: NCT05023759
Title: Anxiety Symptoms in Relation to Use of Hemp-Derived, Full Spectrum Cannabidiol (CBD): a Cohort Study
Brief Title: Anxiety Symptoms in Relation to Use of Hemp-derived, Full Spectrum Cannabidiol (CBD)
Status: Completed | Type: Observational
Sponsor: Formula30A LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: F30A-CBD-GAD2020
Record Dates: First submitted 2021-08-17; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Generalized Anxiety Disorder
Keywords: cannabidiol; endocannabinoid system; CBD; cannabis; anxiety; generalized anxiety disorder; cannabinoids; endocannabinoids; GAD7
MeSH Terms: conditions — Generalized Anxiety Disorder; Marijuana Abuse; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Formula30A Full Spectrum Hemp Cannabidiol 25mg Capsules — Formula30A Full Spectrum Hemp-Derived Cannabidiol (CBD) 25mg Capsules taken once daily for 8 weeks.

SUMMARY:
Generalized anxiety disorder affects about 6.8 million adults in the United States, therefore its treatment is of major public health interest. Cannabidiol (CBD) has shown promise as an effective treatment for anxiety-related symptoms while lacking the severity of adverse effects seen with other medications. Given the wide availability of products containing CBD on the market today, from tinctures to coffee additives, and the undetermined potential for drug-to-drug interactions, medical supervision of CBD intake and formulation-specific clinical research is necessary. Therefore this study aimed to observe the effects of a specific hemp-derived full spectrum CBD formula on anxiety-related symptoms in a group of volunteers. The investigators will examine the self-reported anxiety symptoms in relation to use of a specific CBD formulation (25mg solvent-free full spectrum CBD capsules) in a cohort of adults diagnosed with generalized anxiety disorder. This open-label, cohort study will be conducted at six clinic sites in the United States (including Puerto Rico) from June 2020 through October 2020. The six physicians recruited to participate in the study were each actively prescribing CBD in their practices and were actively caring for patients with anxiety symptoms. Anxiety levels will be measured in enrolled participants diagnosed with generalized anxiety disorder each week for a period of eight weeks using the Generalized Anxiety Disorder 7-Item Scale (GAD7). Participants will also be instructed to take a daily 25mg capsule of CBD. The investigators hypothesize that this formula, when carefully developed and administered by a healthcare professional, will significantly reduce anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 85 years old.
* Research participants of both sexes.
* Good health conditions and without conditions that characterize them as belonging to the risk groups associated with adverse reactions to the product ingredients.
* Research participants with the potential to become pregnant may be included in the study as long as they are sexually abstinent or using a contraceptive method considered effective.
* Signature of the Free and Informed Consent Form.

Exclusion Criteria:

* Initiation of or changes in use of medication or therapies in the past 2 weeks of start of study.
* Pregnancy or breastfeeding.
* History of hepatic compromise with transaminases of 2 times the upper limit of normal or cirrhosis.
* Diagnosis of Bi-Polar disorder, Schizophrenia or Suicidal Ideation.
* Current use of recreational marijuana, medical marijuana, or other CBD formulations.
* History of any substance or alcohol abuse.
* Current use of High Dose or Extended-Release Narcotics.
* Patients diagnosed with sleep apnea.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study conducted at six clinic sites in the United States, primarily Texas and Puerto Rico, from June 2020 through October 2020. Patients with a varying range of anxiety symptoms, who are current patients of the participating clinics and are who diagnosed with generalized anxiety disorder, will be eligible to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 8 weeks | Measured at 8 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.

SECONDARY OUTCOMES:
Participant Clinical Interview with Medical Provider | Measured at 4 weeks after enrollment
Participant Clinical Interview with Medical Provider | Measured at 8 weeks after enrollment

OTHER OUTCOMES:
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 1 week | Measured at 1 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 2 week | Measured at 2 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 3 weeks | Measured at 3 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 4 weeks | Measured at 4 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 5 weeks | Measured at 5 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 6 weeks | Measured at 6 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Change from Baseline Generalized Anxiety Disorder 7-Item Scale (GAD7) Score at 7 weeks | Measured at 7 weeks after baseline
  The Generalized Anxiety Disorder 7-Item (GAD7) score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  The minimum score is 0 and the maximum score is 21, with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - NP Care Clinic, Denton, Texas
  - Dr. Michael Jelinek, MD, Edinburg, Texas
  - Modern Medicine, Forney, Texas
  - Destination Health, Southlake, Texas
  - Melville Medicine, Southlake, Texas
- Dr. Jenaro Velez, MD, Ceiba, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication.
Access Criteria: IPD and additional supporting information shared upon request.

REFERENCES:
- [Background] Skelley JW, Deas CM, Curren Z, Ennis J. Use of cannabidiol in anxiety and anxiety-related disorders. J Am Pharm Assoc (2003). 2020 Jan-Feb;60(1):253-261. doi: 10.1016/j.japh.2019.11.008. Epub 2019 Dec 19. PMID 31866386
- [Background] Blessing EM, Steenkamp MM, Manzanares J, Marmar CR. Cannabidiol as a Potential Treatment for Anxiety Disorders. Neurotherapeutics. 2015 Oct;12(4):825-36. doi: 10.1007/s13311-015-0387-1. PMID 26341731
- [Background] Crippa JA, Derenusson GN, Ferrari TB, Wichert-Ana L, Duran FL, Martin-Santos R, Simoes MV, Bhattacharyya S, Fusar-Poli P, Atakan Z, Santos Filho A, Freitas-Ferrari MC, McGuire PK, Zuardi AW, Busatto GF, Hallak JE. Neural basis of anxiolytic effects of cannabidiol (CBD) in generalized social anxiety disorder: a preliminary report. J Psychopharmacol. 2011 Jan;25(1):121-30. doi: 10.1177/0269881110379283. Epub 2010 Sep 9. PMID 20829306
- [Background] Iffland K, Grotenhermen F. An Update on Safety and Side Effects of Cannabidiol: A Review of Clinical Data and Relevant Animal Studies. Cannabis Cannabinoid Res. 2017 Jun 1;2(1):139-154. doi: 10.1089/can.2016.0034. eCollection 2017. PMID 28861514
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171